CLINICAL TRIAL: NCT05907993
Title: The Effectiveness Of Intravenous Ibuprofen Versus Intravenous Ketorolac For Postoperative Pain Relief After Cesarean Section
Brief Title: Ibuprofen Versus Ketorolac For Postoperative Pain Relief After Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Shehab, MD, lecturer Of Anaesthesia and Surgical intensive care, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0107307
Record Dates: First submitted 2023-04-18; First posted 2023-06-18 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Pain, Postoperative
Keywords: postoperative; pain relief; CESAREAN SECTION
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A): (No Intervention): 30mg ketorolac in 200cc normal saline intravenously every 6hours for 24hours postoperatively.
- Group (B): (Active Comparator): 800mg ibuprofen in 200cc normal saline intravenously every 6 hours for 24hours postoperatively.
  Interventions: Drug: Ibuprofen 800 mg

INTERVENTIONS:
Drug: Ibuprofen 800 mg — Intravenous Ibuprofen versus intravenous Ketorolac for postoperative pain relief
  Arms: Group (B):

SUMMARY:
The aim of this study will be to evaluate the effectiveness of intravenous ibuprofen versus intravenous ketorolac for postoperative pain relief after caesarian section

1. The Primary outcome is measurement of visual analogue score during rest and movement
2. The Secondary outcome is measurement of 24 hours opioids requirements.

DETAILED DESCRIPTION:
METHODS

1. Preoperative assessment:

All parturients included in the study will be assessed thoroughly by:

1. Proper history taking
2. Complete clinical examination.
3. All needed laboratory investigations.

2. Patient preparation:

* On arrival to the operative theatre , an 18 G intravenous cannula will be inserted in a peripheral vein
* Steps of general anaesthesia will be explained to the parturients.

Using a multichannel monitor (mindary) iMeC12 SHENZEN MINDRAY BIO-MEDICAL ELECTRONICS CO, LTD, CHINA, the parturients will be continuously monitored for:

1. Non-invasive arterial blood pressure (NIBP) in (mmHg).
2. Heart rate (beats/min).
3. Oxygen saturation (percentage).
4. End tidal carbon dioxide(mmhg). 3. Anaesthesia technique:

   * Left uterine displacement will be maintained by a wedge under the right hip.
   * Preoxygenation with 100% oxygen will be done for 3-5 minutes
   * For both groups rapid sequence induction will be done with 2mg/kg propofol and 0.9 mg/kg rocuronium,50 microgram fentanyl followed by tracheal intubation and IPPV volume control.
   * Anaesthesia will be maintained with 1.2% isoflurane in 100% Oxygen and 0.1 mg /kg roccuronium will be administrated if needed.
   * After delivery oxytocin infusion 10 IU will be given
   * After finishing operation , inhalational anaesthesia will be stopped and all parturients will receive 2mg/kg sugammadex when train of four is 75%.
   * Then all parturients will be discharged to ward to be put under observation for 24 hours and they will receive NSAID immediately on arrival to the ward .
   * Group A parturients will receive 30 mg ketorolac in 200 cc normal saline intravenously every 6 hours
   * Group B parturients will receive 800 mg Ibuprofen in 200 cc normal saline intravenously every 6 hours
   * All Parturients will receive 25 mg pethidine if visual analogue score (VAS) ≥4.

MEASUREMENTS

The following parameters will be measured for all parturients, in both groups:

1. Demographic data:

   Age (years) Body Mass index ( kilogram/meters2) Weight (kilograms) Height (meters) Duration of surgery (minutes)
2. Postoperative hemodynamics:

   * Heart rate (beats/min)
   * Blood pressure (mmHg)

     1. Baseline value immediately after extubation before giving any analgesia.
     2. Immediately and 2, 4, 6, 12, 24 hours after end of surgery.
3. Visual analogue score:

   * All parturients will be trained to use VAS. VAS at rest (VASR) and during movement (VASM) will be measured at 1,3,6,12,18,24 hours following surgery .The VAS score will be presented as 10 cm horizontal line anchored by the words "no pain"(corresponding to zero) and "worst pain possible"(corresponding to ten).The values will be scored as mild pain(from 1 to 3) ,moderate pain (from 4 to 6) and severe pain (from 7 to 10).
   * If VAS is ≥4 parturients will receive 25mg pethidine iv.
4. Opioid requirement During the first 24 hours after surgery(mg) The doses of pethidine required during the first 24 hours postoperatively will be calculated.
5. Nocturnal awakening due to pain (percentage) The percentage of parturients who become awake at night due to pain
6. Time to ambulate (minutes) The time the parturient takes to get out of bed and to do light activities such as sitting, standing or walking.
7. Time to first analgesic dose (minutes) rescue analgesia The time when the patient require the first analgesic dose in the ward.

ELIGIBILITY:
Inclusion Criteria:

1. Parturients aged 20-30years.
2. ASA physical satatus: II.
3. Anticipated hospital stay for at least 24 hours.
4. Refusal of spinal anaesthesia.

Exclusion Criteria:

1. Known allergy to the used drugs.
2. Renal and hepatic impairement
3. History of brochial asthma.
4. Low platelets count (<70000).
5. Bleeding diathesis and with history or risk of intracranial hemorrhage.
6. Obese and morbidly obese parturients.
7. GIT problems as gastritis or GI bleeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant Females
Enrollment: 50 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
measurement of visual analogue score | after the surgery average 24 hours postoperative
  measurement of visual analogue score during rest and movement . The Score range from 0- 10 . 0 means no pain and 10 indicates the worst pain ever

SECONDARY OUTCOMES:
opioids requirements. | after the surgery average 24 hours postoperative
  Total opioid cumulative requirement dose

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S. Shehab, MD, Principal Investigator — Alexandria University
Locations (1):
- Ahmed S. Shehab, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
17. there is a plan to make individual participant data (IPD) collected in this study, including data dictionaries, available to other researchers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: to the time when summary data are published
Access Criteria: Accessible through the web site

REFERENCES:
- [Background] Ekinci M, Ciftci B, Celik EC, Kose EA, Karakaya MA, Ozdenkaya Y. A Randomized, Placebo-Controlled, Double-Blind Study that Evaluates Efficacy of Intravenous Ibuprofen and Acetaminophen for Postoperative Pain Treatment Following Laparoscopic Cholecystectomy Surgery. J Gastrointest Surg. 2020 Apr;24(4):780-785. doi: 10.1007/s11605-019-04220-1. Epub 2019 Apr 22. PMID 31012040
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31012040/